CLINICAL TRIAL: NCT01629810
Title: An Unblinded Crossover Study of The Use of Whole-Body Periodic Acceleration Therapy To Treat Pain, Stiffness, Abnormal Gait and Balance
Brief Title: Use of Whole-Body Periodic Acceleration Therapy To Aches and Pains
Acronym: Exer-Rest
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Translational Medicine (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20110957
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Pain; Stiffness; Abnormal Gait; Balance
Keywords: Motion platform at appropriate settings.; Relief of pain.; Improvement in quality of life, cognition, and mood.; Effects of WBPA on cognition, mood, behavior, and functioning.; Dose response effect .; Gather data for long-term (2 year) study
MeSH Terms: conditions — Pain; Mobility Limitation; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Whole body periodic acceleration (Exer-Rest) — Lying on the vibrating bed for 45 minutes per session for 10 sessions over 2 weeks.

SUMMARY:
The purpose of this study is to test the effectiveness of whole body periodic acceleration for helping with symptoms of aches and pains suffered by many patients.

DETAILED DESCRIPTION:
This is an unblinded cross-over study of whole-body periodic acceleration (WBPA) to ascertain if this treatment modality provides symptomatic relief of pain, stiffness, and abnormal gait and balance in a variety of conditions. The study will compare a specific mechanism of motion, whole-body periodic acceleration (WBPA), that has been shown to increase the release of beneficial mediators from the vascular endothelium into the circulation, to a control condition of slow passive motion that promotes relaxation but does not increase release of beneficial mediators into the circulation. The study tests the efficacy and safety of a commercially available device that consists of a motion platform, called Exer-Rest©, that is capable of producing both types of motion to be tested. In this investigation, 15 subjects will be randomly assigned to either procedure for 10 treatments for 2 weeks followed by a one-week "wash-out" period. Then the opposite treatment will be employed for two weeks.

ELIGIBILITY:
Inclusion Criteria:

Subjects qualifying for this study satisfy the following criteria:

1. Over 18 years of age;
2. Complain of either chronic pain, joint stiffness, and/or dysfunctions of gait and balance;
3. Complaints have been annotated by a competent physician, and the subject has been evaluated for conditions that commonly contribute to the respective symptoms;
4. Capable of completing the appropriate testing and baseline assessments, such as quantitative electroencephalography (qEEG) and questionnaires;
5. Tolerate the motion and duration of treatment of the WBPA.
6. Be available for regular visits to the research site for the duration of the study.

Exclusion Criteria:

WBPA is contraindicated for subjects who are pregnant or who suffer with unexplained leg pain, skin eruptions, or who have unstable spinal injuries or conditions. Subjects who cannot tolerate the motion and duration of treatment are also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Self-report of pain | 2 weeks
  Self-report of pain at start and completion of first course of treatment lasting for 2 weeks.

SECONDARY OUTCOMES:
Quality of life | 2 weeks
  Self-report of change in quality following 2 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Translational Medicine Group, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sackner MA, Gummels E, Adams JA. Effect of moderate-intensity exercise, whole-body periodic acceleration, and passive cycling on nitric oxide release into circulation. Chest. 2005 Oct;128(4):2794-803. doi: 10.1378/chest.128.4.2794. PMID 16236957